CLINICAL TRIAL: NCT05071183
Title: A Phase 1b/2 Study of Repotrectinib in Combination With Other Anticancer Therapies for the Treatment of Subjects With KRAS-Mutant Advanced Solid Tumors (TRIDENT-2)
Brief Title: A Study of Repotrectinib in Combination With Other Anticancer Therapies for the Treatment of Subjects With KRAS-Mutant Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Inability to achieve and optimize a dose that could provide a positive benefit risk profile
Sponsor: Turning Point Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA127-1025; CA127-1025 (Other: BMS Protocol ID); TPX-0005-13 (Other: Turning Point Therapeutics Protocol ID)
Expanded Access: NCT05926232 (Available)
Record Dates: First submitted 2021-09-13; First posted 2021-10-08 (Actual); Results first posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: KRAS Mutation-Related Tumors; Metastatic Solid Tumor; Advanced Solid Tumor
Keywords: KRAS; KRAS-mutant; Metastatic Solid Tumor; Advanced Solid Tumor; Advanced/metastatic disease
MeSH Terms: conditions — Neoplasm Metastasis | interventions — repotrectinib; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TPX-0005 + Trametinib (Experimental): TPX-0005 + Trametinib Dose Escalation and Dose Expansion
  Dose escalation: KRAS G12D mutant advanced solid tumors. Dose expansion: KRAS G12D locally advanced or metastatic NSCLC
  Interventions: Drug: TPX-0005; Drug: Trametinib

INTERVENTIONS:
Drug: TPX-0005 — Oral TPX-0005 capsules
  Other Names: repotrectinib
Drug: Trametinib — Oral trametinib tablets
  Other Names: Mekinist

SUMMARY:
A Phase 1b/2 Study of Repotrectinib in Combination with Other Anticancer Therapies for the Treatment of Subjects with KRAS-Mutant Advanced Solid Tumors (TRIDENT-2)

DETAILED DESCRIPTION:
Phase 1 Dose Escalation: To evaluate tolerability of repotrectinib at increasing dose levels in combination with other anticancer therapies for the treatment of subjects with locally advanced or metastatic KRAS-mutant solid tumors

Phase 2 Efficacy Evaluation: Investigate the anti-tumor efficacy and safety of repotrectinib in combination with other anticancer therapies for the treatment of patients with locally advanced or metastatic KRAS-mutant solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 (or as required by local regulation).
* Histological or cytological confirmation of unresectable or metastatic solid tumor malignancy harboring a KRAS mutation.
* No more than 3 prior standard treatments appropriate for tumor type and stage of disease.
* ECOG performance status ≤ 1.
* Existence of measurable disease (according to Response evaluation criteria in solid tumors [RECIST v1.1] criteria).
* Subjects with asymptomatic CNS metastases and/or asymptomatic leptomeningeal carcinomatosis are eligible.
* Adequate organ function.

Exclusion Criteria:

* Major surgery within four weeks of the start of treatment.
* Previous other cancer requiring treatment within the previous two years.
* Clinically significant cardiovascular disease.
* Any of the following cardiac criteria:
* Mean resting corrected QT interval (QTc) > 470 msec obtained from three ECGs and any factors that increase the risk of QTc prolongation or arrhythmic events
* Any clinically important abnormalities in rhythm, conduction, or morphology of resting ECG
* Known clinically significant active infections not controlled with systemic treatment (bacterial, fungal, viral including HIV positivity).
* Gastrointestinal disease or other malabsorption syndromes that would impact drug absorption.
* Subjects being treated with or anticipating the need for treatment with strong CYP3A inhibitors or inducers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-09-23 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (6):
- United States (6):
  - Local Institution - 2101, California City, California
  - Local Institution - 2109, California City, California
  - Local Institution - 2106, Denver, Colorado
  - Local Institution - 2108, Nashville, Tennessee
  - Local Institution - 2107, Houston, Texas
  - Local Institution - 2102, Virginia Beach, Virginia

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSStudyConnect.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 9 participants enrolled and treated in phase 1. No participants enrolled in phase 2.
Groups:
- Dose Level 1: Repotrectinib 120 mg QD, Trametinib 2 mg QD
- Dose Level 2: Repotrectinib 120 mg QD, Trametinib 1.0 mg QD
- Dose Level -2a: Repotrectinib 160 mg QD, Trametinib 1.0 mg QD
Period: Overall Study
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level -2a
Started | 2 | 5 | 2
Completed | 0 | 0 | 0
Not Completed | 2 | 5 | 2
Not completed — Death | 1 | 2 | 0
Not completed — Other Reasons | 1 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level -2a | Total
Number analyzed (Participants) | 2 | 5 | 2 | 9
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.5 (21.92) | 61.8 (12.74) | 60.5 (13.44) | 61.0 (12.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 1 | 7
  Male | 0 | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 3 | 2 | 7
  Unknown or Not Reported | 0 | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 0 | 5 | 1 | 6
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities
Description: Number of participants with first cycle DLTs to determine Mean Tolderable Dose (MTD) and/or RP2D.
  A DLT is defined as an adverse event (AE) or abnormal laboratory value assessed as unrelated to disease progression, intercurrent illness, or concomitant medications that meets the criteria defined in each subprotocol.
  The MTD is defined as the highest dose level of repotrectinib given in combination with other anticancer therapy observed to cause a DLT in fewer than 33% of the treated subjects in the first treatment cycle (i.e., Cycle 1).
Time Frame: From initial dose to end of first cycle of treatment, approximately 28 days
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level -2a
Number analyzed (Participants) | 2 | 5 | 2
Participants | 2 | 0 | 2

2. Secondary Outcome: Overall Response Rate (ORR) Assessed the Investigator Using RECIST v1.1.
Description: The ORR will be defined as the percentage of participants with a confirmed complete response (CR) or partial response (PR). A confirmed response is a response that persists on a repeat imaging performed at least 4 weeks after initial documentation of response. Participants with a confirmed objective response (CR or PR) will be referred to as responders.
  Radiographic confirmation of objective tumor response (CR or PR) or disease progression will be based on RECIST v1.1. The ORR will be reported as the percentage of responders by RECIST v1.1 along with the corresponding two-sided 95% Clopper-Pearson exact CI.
  Complete Response (CR) = Disappearance of all target lesions Partial Response (PR) = >=30% decrease in the sum diameters of target lesions.
Time Frame: From screening to end of treatment approximately 10 months
Population: Efficacy Evaluable Set - all participants who (1) received at least one dose of study treatment with repotrectinib; (2) KRAS mutation determined by a qPCR or NGS test performed in a CLIA laboratory or equivalently accredited diagnostic lab; (3) have a baseline tumor assessment with measurable disease and have at least 1 on-study tumor assessment per RECIST v1.1; and (4) have no major protocol violations that could affect efficacy. (Dose Level 1 and -2a did not meet efficacy evaluable criteria)
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level -2a
Number analyzed (Participants) | 0 | 4 | 0
Percentage of Participants |  | 0 [0.0 to 60.2] |

3. Secondary Outcome: Cmax of Repotrectinib
Description: Cmax is defined as maximum plasma concentration of the drug.
Time Frame: At Cycle 1 Day 1 and Cycle 1 Day 22
Population: All Treated Participants with evaluable pharmacokinetic measurements.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level -2a
Number analyzed (Participants) | 2 | 5 | 2
ng/mL
  Cycle 1 Day 1 | 656.85 (37.88) | 570.86 (66.02) | 569.27 (20.26)
  Cycle 1 Day 22: number analyzed (Participants) | 0 | 2 | 0
  Cycle 1 Day 22 |  | 411.83 (49.37) |

4. Secondary Outcome: Tmax of Repotrecitinib
Description: Tmax is defined is the time to maximum plasma concentration
Time Frame: At Cycle 1 Day 1 and Cycle 1 Day 22
Population: All Treated Participants with evaluable pharmacokinetic measurements.
Measure: Median (Full Range); unit: hours (h)
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level -2a
Number analyzed (Participants) | 2 | 5 | 2
hours (h)
  Cycle 1 Day 1 | 3.00 [2.00 to 4.00] | 2.00 [1.00 to 6.00] | 4.00 [4.00 to 4.00]
  Cycle 1 Day 22: number analyzed (Participants) | 0 | 2 | 0
  Cycle 1 Day 22 |  | 3.00 [2.00 to 4.00] |

5. Secondary Outcome: AUC 0-24 of Repotrecitinib
Description: Area under the plasma concentration time-curve. AUC from time 0 to 24 hours after dose.
Time Frame: At Cycle 1 Day 1 and Cycle 1 Day 22
Population: All Treated Participants with evaluable pharmacokinetic measurements.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level -2a
Number analyzed (Participants) | 2 | 5 | 2
h*ng/mL
  Cycle 1 Day 1 | 6208.74 (82.59) | 6692.13 (57.48) | 8327.26 (25.27)
  Cycle 1 Day 22: number analyzed (Participants) | 0 | 2 | 0
  Cycle 1 Day 22 |  | 5223.89 (31.06) |

6. Secondary Outcome: Cmax of Trametinib
Description: Cmax is defined as maximum plasma concentration of the drug.
Time Frame: At Cycle 1 Day 1 and Cycle 1 Day 22
Population: All Treated Participants with evaluable pharmacokinetic measurements.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level -2a
Number analyzed (Participants) | 2 | 5 | 2
ng/mL
  Cycle 1 Day 1 | 15.24 (20.55) | 3.30 (69.58) | 2.60 (29.74)
  Cycle 1 Day 22: number analyzed (Participants) | 0 | 2 | 0
  Cycle 1 Day 22 |  | 10.55 (56.36) |

7. Secondary Outcome: Tmax of Trametinib
Description: Tmax is defined is the time to maximum plasma concentration
Time Frame: At Cycle 1 Day 1 and Cycle 1 Day 22
Population: All Treated Participants with evaluable pharmacokinetic measurements.
Measure: Median (Full Range); unit: hours (h)
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level -2a
Number analyzed (Participants) | 2 | 5 | 2
hours (h)
  Cycle 1 Day 1 | 1.50 [1.00 to 2.00] | 2.00 [1.00 to 2.00] | 2.00 [2.00 to 2.00]
  Cycle 1 Day 22: number analyzed (Participants) | 0 | 2 | 0
  Cycle 1 Day 22 |  | 2.50 [1.00 to 4.00] |

8. Secondary Outcome: AUC 0-24 of Trametinib
Description: Area under the plasma concentration time-curve. AUC from time 0 to 24 hours after dose.
Time Frame: At Cycle 1 Day 1 and Cycle 1 Day 22
Population: All Treated Participants with evaluable pharmacokinetic measurements.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level -2a
Number analyzed (Participants) | 2 | 5 | 2
h*ng/mL
  Cycle 1 Day 1 | 88.77 (6.48) | 20.58 (36.19) | 19.27 (13.47)
  Cycle 1 Day 22: number analyzed (Participants) | 0 | 2 | 0
  Cycle 1 Day 22 |  | 197.45 (45.52) |

ADVERSE EVENTS:
Time Frame: From first dose to 28 days after last dose, approximately 9.5 months
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants.
  The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level -2a
All-Cause Mortality (participants affected / at risk) | 2/2 | 2/5 | 1/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 1/5 | 2/2
Other Adverse Events (participants affected / at risk) | 2/2 | 5/5 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 (N=2) | Dose Level 2 (N=5) | Dose Level -2a (N=2)
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 (N=2) | Dose Level 2 (N=5) | Dose Level -2a (N=2)
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Periorbital oedema (Eye disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 2 | 1
Paraesthesia oral (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2 | 1
Asthenia (General disorders) | 0 | 2 | 1
Catheter site oedema (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 1 | 2 | 1
Gait disturbance (General disorders) | 0 | 1 | 0
COVID-19 (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Amylase increased (Investigations) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0
Lipase increased (Investigations) | 0 | 0 | 1
White blood cell count increased (Investigations) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Aphasia (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 2 | 1
Dysgeusia (Nervous system disorders) | 0 | 2 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0
Euphoric mood (Psychiatric disorders) | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Embolism (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Study terminated early by sponsor before initiation of phase 2, so phase 2 outcome measures and endpoint data will not be reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-04): https://cdn.clinicaltrials.gov/large-docs/83/NCT05071183/Prot_SAP_000.pdf